CLINICAL TRIAL: NCT06742827
Title: Effectiveness of an Educational Intervention by Nurses Supported by ICTs to Improve Therapeutic Adherence in People Undergoing Hemodialysis Treatment
Brief Title: Educational Intervention and Adherence
Acronym: Hemodialysis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEI-FE 2024-136
Record Dates: First submitted 2024-12-04; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Treatment Adherence and Compliance; Effectiveness; Renal Dialysis; Nurse's Role
Keywords: Treatment Adherence and Compliance; Effectiveness; Renal Dialysis; Nursing
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention group: participants will receive an educational intervention on hemodialysis adherence)
  Interventions: Other: educational intervention based on information and communication technologies.
- Control (No Intervention): Control group:participants will receive conventional care provided by health professionals

INTERVENTIONS:
Other: educational intervention based on information and communication technologies. — will be carried out through a mobile application, which will be installed on each person's device, as well as short text messages will be sent and counseling will be available 24/7. The contents of the application will be educational and will be elaborated framed in the following components: understanding of the disease and the consequences of not adhering (comprehensibility) to the treatment, maintaining a balance between the psychosocial resources that the patient has and the demands that the disease places on them (manageability), and the involvement of the person in decision making and the sense of continuing to adhere to hemodialysis treatment (meaningfulness).
  Other Names: ICT educational intervention
  Arms: Intervention

SUMMARY:
quasi-experimental, parallel study, with the objective of evaluating the effectiveness of an educational nursing intervention supported by ICTs, for the improvement of therapeutic adherence in people undergoing hemodialysis treatment in a renal unit in Barranquilla (Colombia)

DETAILED DESCRIPTION:
This study is quantitative in approach and will be conducted in three phases: Phase I: development of the intervention, Phase II: validation by expert consensus for the content of the nursing intervention. Phase III a randomized clinical trial.

I. Development of the intervention During this phase knowledge gained from theoretical and empirical approaches will play a key role in creating an effective intervention aimed at improving treatment adherence in hemodialysis patients. An intervention guided by salutogenic theory and mediated by ICTs will be used. Each of these approaches provides a unique and valuable perspective that enriches our understanding of the problem, thus facilitating informed decision making during the planning and implementation phase of interventions.

As for the theoretical-empirical understanding of the problem, which will perform the combination of theoretical and empirical approach in order to make the clear identification of the problem, requiring resolution of its determinants, severity, consequences, as well as, evidencing the support of the intervention through the incorporation of theories that guide the development of the intervention while seeking to establish the relationship between the characteristics of the problem and empirical components.

Description of the Nursing Educational Intervention:

Regarding the theoretical approach, Antonovsky's salutogenic theory is incorporated, which makes it possible to understand the problem. This theory, which is broad and comprehensive, adopts a salutogenic perspective by viewing people as biopsychosocial beings who make choices in their lives. It allows individuals to identify the psychosocial resources that contribute to maintaining their health and well-being. In this sense, Antonovsky introduces the concept of "sense of coherence", which comprises the elements of comprehensibility (knowledge), manageability (behavior) and meaningfulness (motivation).

From the empirical approach, the literature review has revealed that therapeutic adherence is a complex phenomenon, influenced by a variety of factors and has been the subject of study in various disciplines, including nursing. To address this issue effectively, it is necessary to implement educational interventions that promote health and well-being in people undergoing hemodialysis.

Content of the Intervention:

Regarding delivery strategies, it will be carried out through a mobile application, which will be installed on each person's device, likewise short text messages will be sent and counseling will be done with 24/7 counseling availability. The contents of the application will be educational and will be developed within the framework of the following components

II. RANDOMIZED CLINICAL TRIAL:

Type of study. Intervention study of the parallel type randomized controlled clinical trial type. For the reporting of the results, the extent of the Consort Statement for randomized clinical trials of non-pharmacological interventions will be taken into account. The randomized controlled trial is considered to be the most rigorous and robust research method for determining whether a cause-effect relationship exists between an intervention and an outcome.

Study Setting. The study will be carried out in a renal unit in the city of Barranquilla.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old
* In hemodialysis treatment for at least 3 months for three or four hours, with a frequency of three times a week in a renal
* Must live in Barranquilla
* Must be independent in self-care activities such as being able to walk and eat without assistance
* Must have access to an Android or Apple cell phone which is in daily use.

Exclusion Criteria:

* Signs or symptoms as a result of target organ damage
* Cognitive, hearing or visual impairments that prevent them from adequately receiving the educational intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Score of ESRD-AQ | PRE (baseline, pre-intervention) and POST (immediately after the intervention)
  Score of the End-Stage Renal Disease-Adherence Questionnaire (ESRD-AQ)
Score of SOC | PRE (baseline, pre-intervention) and POST (immediately after the intervention)
  Score of the scale Sense of Coherence (SOC)

CONTACTS AND LOCATIONS:
Locations (1):
- Barranquilla, Barranquilla, Atlántico, Colombia

REFERENCES:
- [Background] Park J, Park J. Identifying the Knowledge Structure and Trends of Nursing Informatics: A Text Network Analysis. Comput Inform Nurs. 2023 Jan 1;41(1):8-17. doi: 10.1097/CIN.0000000000000919. PMID 35703232
- [Background] Newman MA, Smith MC, Pharris MD, Jones D. The focus of the discipline revisited. ANS Adv Nurs Sci. 2008 Jan-Mar;31(1):E16-27. doi: 10.1097/01.ANS.0000311533.65941.f1. No abstract available. PMID 20531258
- [Background] Goode CJ. Evaluation of research-based nursing practice. Nurs Clin North Am. 1995 Sep;30(3):421-8. PMID 7567568
- [Background] Mittelmark MB, Bull T. The salutogenic model of health in health promotion research. Glob Health Promot. 2013 Jun;20(2):30-8. doi: 10.1177/1757975913486684. PMID 23797938
- [Background] Arad M, Goli R, Parizad N, Vahabzadeh D, Baghaei R. Do the patient education program and nurse-led telephone follow-up improve treatment adherence in hemodialysis patients? A randomized controlled trial. BMC Nephrol. 2021 Apr 7;22(1):119. doi: 10.1186/s12882-021-02319-9. PMID 33827478
- [Background] Banning M. A review of interventions used to improve adherence to medication in older people. Int J Nurs Stud. 2009 Nov;46(11):1505-15. doi: 10.1016/j.ijnurstu.2009.03.011. Epub 2009 Apr 24. PMID 19394018